CLINICAL TRIAL: NCT03936699
Title: Safety and Effectiveness of Transcutaneous Electrical Nerve Stimulation (TENS)-Assisted Weight Loss and/or Appetite Suppression
Brief Title: ELIRA 2: Safety and Effectiveness of TENS Assisted Weight Loss and Appetite Suppression
Acronym: ELIRA_2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Elira Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CD-005
Record Dates: First submitted 2018-06-29; First posted 2019-05-03 (Actual); Results first posted 2022-02-02 (Actual); Last update posted 2022-02-02 (Actual); Status verified 2021-12

CONDITIONS: Weight Loss
MeSH Terms: conditions — Weight Loss | interventions — Diet; Exercise

STUDY DESIGN:
Intervention Model Description: Randomized, adaptive parallel arm study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Treatment (Experimental): The Transcutaneous Nerve Stimulator (TENS) Elira wearable patch system will be applied to varying locations on the T6/T7 dermatome for 30 minutes three times a day after meals. Subjects will be instructed to follow a 1200 calorie healthy diet and record any changes in appetite.
  Interventions: Device: Transcutaneous Nerve Stimulator (TENS); Behavioral: Diet & Exercise
- Control (Active Comparator): Open label diet and exercise counseling only. Subjects will be instructed to follow a healthy 1200 calorie diet and record any changes in appetite.
  Interventions: Behavioral: Diet & Exercise

INTERVENTIONS:
Device: Transcutaneous Nerve Stimulator (TENS) — The Elira wearable patch system is a Radio Frequency (RF) coupled, wearable transcutaneous electrical nerve stimulator (TENS) device controlled via Bluetooth by a smart phone unit running a custom application which directs therapy from the patch within safe limits set by a clinician and also includes a weight loss diary.
  Behavioral: Diet & Exercise Subjects to be instructed on a healthy 1200 calorie diet.
  Arms: Treatment
Behavioral: Diet & Exercise — Subjects to be instructed on a healthy 1200 calorie diet.

SUMMARY:
The objectives of this study are to demonstrate safety and effectiveness of a wearable patch TENS system (Appendix 2) in driving weight loss and appetite suppression when coupled with an integrated weight loss reduction strategy. The study is designed to demonstrate that TENS stimulation sufficient to drive weight loss and appetite suppression is safe and tolerable when compared to standard of care, and that adverse events/adverse device effects are similar to other TENS device use cases.

DETAILED DESCRIPTION:
Randomized, adaptive parallel arm study. Subjects will be initially screened during a screening period (+/- 7 days). During this screening period, subjects will sign an Informed Consent Form (ICF), have their weight/height and blood pressure measured as part of a physical exam, take a pregnancy test (females of child bearing potential), get blood drawn for analysis (blood lipids, HbA1c), and complete the PHQ-9 and pre-study survey.

At the end of the screening period, eligible subjects will be enrolled/randomized in the study and be randomized to either a treatment or control group. After enrolling, both control and treatment subjects will be instructed to follow a healthy diet and reduce calories as desired for the duration of the study and will receive training on the use of the electronic scale and completion of paper diaries. For the treatment group, subjects will be instructed on use of the Elira wearable patch system. Photographs will be taken at the enrollment visit. Following this, subjects will enter the Therapy Period for ~24-weeks.

At the 12 week visit, subjects will be assessed for weight loss, blood pressure, blood lipids, HbA1c, patient preference questionnaire and their participation will continue through months 4-6 for the Safety phase of the Therapy Period. The Therapy Period will be considered complete (pending laboratory results, adverse events or serious adverse events). Patient (treatment) photographs will also be taken at the 12 week visit.

The study utilizes an adaptive approach where cohorts of enrolled/randomized subjects (in groups of ~25 per arm) are assessed for dose response and progression to achievement of primary and secondary endpoints. Frequent interim endpoint assessment utilizing Markov-chain Monte Carlo (MCMC) methods coupled with Longitudinal analyses will be utilized to determine sample sizes for future cohorts (assessed primarily via Normal dynamic linear modeling [NDLM]). Long term safety of the device will be shown through 6 months of usage.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is between 18 - 65 years of age inclusive.
2. Subject has a BMI of 25-35 kg/ m2 inclusive.
3. Subject has signed the informed consent form and is able to comply with study protocol and adhere to study visit schedule.
4. Subject is able to wear and use a wearable, patch TENS system.
5. Subject is able to use a touch screen hand held smart phone.
6. Subject is fluent in English and can complete questionnaires.
7. Females of childbearing potential (FOCBP) must have a negative urine pregnancy test at screening or enrollment visit, prior to placement of ELIRA device.
8. Subject is male or non-pregnant, non-lactating female, who agrees to use effective contraceptive methods throughout the length of the trial based on PI approval.

Exclusion Criteria:

1. Subject has any known gastrointestinal disorder that in the opinion of the PI precludes enrollment into the trial.
2. Subject has had a prior bariatric procedure or any previous procedure on the stomach.
3. Subject has any significant multisystem disease in the opinion of the PI.
4. Subject has > 6.5 HbA1c.
5. Subject has significant cardiac arrhythmia, ectopy, or significant cardiovascular disease.
6. Subject has an existing implanted electrical stimulator (e.g., pacemaker, AICD).
7. Subject is a female of child-bearing potential who is pregnant or intends to become pregnant during the trial period.
8. Subject has current and/or a history of cancer within the past 5 years (not including basal cell carcinoma or cervical carcinoma in situ).
9. Subject has had a weight change of + 5% of his/her Total Body Weight in the 3 months prior to screening.
10. Subject has a moderate / severe psychiatric disorder.
11. Subject has a diagnosed neurological disease.
12. Subject has a diagnosed eating disorder.
13. Subject has a skin disorder affecting the thoracic dermatomes.
14. Subject has active or /has ever had shingles in the abdominal area.
15. Subject has abdominal surgery or other scars which may interfere with TENS stimulation in the opinion of the PI.
16. Subject is currently enrolled in other potentially confounding research.
17. Subject has known allergic reaction to materials in the TENS electrodes and/or is otherwise unable to tolerate stimulation with the wearable TENS system. This includes known allergies to latex, nickel and/or hydrogels.
18. Subject has a history of sensitive skin, including eczema wheel-and-flare or other skin irritation, per PI discretion.
19. Subject is actively participating or unwilling to discontinue participation in another weight loss program. Subjects may not enroll in paid or unpaid programs that involve in-person or online apps or coaching, beginning new fitness regimens or utilizing meal planning or paid nutritional coaching during the course of the ELIRA study
20. Subject is taking weight loss control medications including but not limited to Over The Counter (OTC) medications, Metformin, and Belviq. (See Appendix 8)
21. Subject is planning any major medical treatments or surgeries that could cause weight loss.
22. Subject is unable to take anti-nausea medications planned for the study.
23. Inability to walk at least 0.8 kilometers per day (10 minutes of continuous walking).
24. Current smoker or user of nicotine product or smoking cessation within 1 year of the screening date.
25. History of treatment for or current abuse of drug or alcohol.
26. A score of ≥10 on the Patient Health Questionnaire 9 (PHQ-9), demonstrating moderate depression.
27. Any subject that the investigator considers inappropriate for the study for medical reasons.
28. Subject has a history of moderate/severe migraines or other severe headache disorders requiring the treatment of Topiramate.
29. Subject is on drug therapy which may alter antral motility or appetite, per PI discretion.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2018-06-22 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2019-05-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- West County OB/GYN Specialists, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment: The Transcutaneous Nerve Stimulator (TENS) Elira wearable patch system will be applied to varying locations on the T6/T7 dermatome for 30 minutes three times a day after meals. Subjects will be instructed to follow a 1200 calorie healthy diet and record any changes in appetite.
  Transcutaneous Nerve Stimulator (TENS): The Elira wearable patch system is a Radio Frequency (RF) coupled, wearable transcutaneous electrical nerve stimulator (TENS) device controlled via Bluetooth by a smart phone unit running a custom application which directs therapy from the patch within safe limits set by a clinician and also includes a weight loss diary.
  Behavioral: Diet & Exercise Subjects to be instructed on a healthy 1200 calorie diet.
  Diet & Exercise: Subjects to be instructed on a healthy 1200 calorie diet.
Period: Overall Study
Arm/Group | Treatment | Control
Started | 83 | 78
Completed | 61 | 55
Not Completed | 22 | 23

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment | Control | Total
Number analyzed (Participants) | 83 | 78 | 161
Age, Continuous [Mean (Full Range); unit: years] | 48 [26 to 65] | 48 [25 to 64] | 48 [25 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77 | 73 | 150
  Male | 6 | 5 | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White, non-Hispanic | 69 | 66 | 135
  Black | 9 | 9 | 18
  Asian | 2 | 1 | 3
  Other | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  United States | 83 | 78 | 161
BMI [Mean (Full Range); unit: kg/m^2] | 31.6 [25.1 to 36.3] | 31.5 [25.2 to 36.5] | 31.6 [25.1 to 36.5]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events
Description: Treatment Emergent Adverse Events [Time Frame: 12 weeks] Safety/Tolerability will be assessed by the non-inferiority of incidence of serious adverse events (SAEs), unanticipated serious adverse events (USAEs), device-related SAEs (DSAEs), and unanticipated device-related SAEs (UDAEs) that are associated with the TENS therapy throughout the stimulation and the follow-up period versus historical control (compared with other TENS systems).
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Control
Number analyzed (Participants) | 61 | 55
Participants | 0 | 0

2. Primary Outcome: Change in Appetite as Measured by a Visual Analogue Scale From Baseline
Description: Appetite Changes [Time Frame: 12 weeks] Percent change in appetite scores at the end of the trial compared to Baseline between Treatment and Control.
  Subjects are asked to score level of satisfaction, fullness, hunger and ability to eat on a Visual Analogue Scale of 1 to 100 before and after meals with lower scores indicating lower satisfaction, fullness, hunger or ability to eat, respectively. Scores are captured in a diary once a week with 8 time points. The weeks are captured as week 0 through week 12. The time points at each week include:
  * 30 minutes before breakfast
  * 30, 60, and 90 minutes after breakfast
  * Pre-lunch
  * Midafternoon
  * 30 minutes before dinner
  * Bedtime For each of the four appetite suppression variables (satisfaction, fullness, hunger and ability to eat), the 8 time points at week zero will be averaged for the baseline score (baseline), and the 8 time points at week 12 will be averaged for the 3-month score (3month).
Time Frame: 3 months
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of change
Arm/Group | Treatment | Control
Number analyzed (Participants) | 71 | 65
percentage of change
  VAS Satisfaction | -4.1 [-16.4 to 8.1] | 16.6 [3.8 to 29.3]
  VAS Fullness | 36.6 [24 to 49.3] | 10.9 [-2.3 to 24.2]
  VAS Hunger | 28.2 [18 to 38.4] | 8.2 [-2.5 to 18.8]
  VAS Amount Able to Eat | -15 [-22.7 to -7.3] | 7.7 [-0.4 to 15.8]

3. Secondary Outcome: Change in Percent Total Body Weight Loss
Description: Percent reduction in total body weight loss (%TBWL), measured as End Weight - Initial Weight, multiplied by 100, at the end of Experimental period compared to Baseline between Treatment and Control.
Time Frame: 3 months
Measure: Mean (Full Range); unit: percent total body weight loss
Arm/Group | Treatment | Control
Number analyzed (Participants) | 63 | 59
percent total body weight loss | -2.56 [-11.88 to 6.4] | -1.09 [-12.59 to 4.77]

4. Secondary Outcome: Changes in BMI
Description: Changes in BMI [ Time Frame: 3 months ]
Time Frame: 3 months
Measure: Mean (Full Range); unit: kg/m^2
Arm/Group | Treatment | Control
Number analyzed (Participants) | 63 | 59
kg/m^2 | 0.79 [-3.21 to 5.76] | 0.14 [-3.55 to 4.29]

ADVERSE EVENTS:
Time Frame: Adverse Events [Time Frame: 12 weeks]
Arm/Group | Treatment | Control
All-Cause Mortality (participants affected / at risk) | 0/83 | 0/78
Serious Adverse Events (participants affected / at risk) | 0/83 | 0/78
Other Adverse Events (participants affected / at risk) | 55/83 | 23/78
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=83) | Control (N=78)
Rash, Hives (Skin and subcutaneous tissue disorders) | 15 (15) | 2 (2)
Atypical chest pain (Cardiac disorders) | 0 (0) | 1 (1)
Heartburn (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal cramping / stomach pain (Gastrointestinal disorders) | 4 (4) | 0 (0)
Back spasms / pain / cramping (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Bruise on abdomen (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Carpal tunnel repair (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Flu (Infections and infestations) | 1 (1) | 1 (1)
Gastroenteritis (Gastrointestinal disorders) | 2 (2) | 1 (1)
Hypothyroidism (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Left foot injury (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Plantar fascitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Posterior tibial tendon insufficiency (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Stomach flu (Infections and infestations) | 0 (0) | 1 (1)
Tooth pain (General disorders) | 0 (0) | 1 (1)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 6 (6)
Urinary tract infection (Renal and urinary disorders) | 1 (1) | 2 (2)
Broken ankle / fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 1 (1)
Bunion surgery (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Gout (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Loose stools (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hip pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Sciatica (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Shingles (Infections and infestations) | 3 (3) | 0 (0)
Slipped disc / back injury (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Toe fungus (Infections and infestations) | 1 (1) | 0 (0)
Shoulder pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cholelithitis (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-03): https://cdn.clinicaltrials.gov/large-docs/99/NCT03936699/Prot_SAP_001.pdf